CLINICAL TRIAL: NCT07009717
Title: The Role Of Great Toe Strength And Its Association With The Severity Of Symptoms Of Chemotherapy-Induced Peripheral Neuropathy (CIPN)
Brief Title: Relationship Between Great Toe Strength And Symptoms of Chemotherapy-Induced Peripheral Neuropathy (CIPN)
Status: Recruiting | Type: Observational
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Other Study IDs: IRB202401631
Record Dates: First submitted 2025-05-29; First posted 2025-06-08 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2025-08

CONDITIONS: Chemotherapy-induced Peripheral Neuropathy (CIPN); Healthy
Keywords: Great Toe strength; chemotherapy-induced peripheral neuropathy; muscle weakness; clinical biomarker; force development curve
MeSH Terms: conditions — Muscle Weakness | interventions — Observation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CIPN: Individuals with chemotherapy-induced peripheral neuropathy with a confirmed diagnosis using the nerve conduction study
  Interventions: Other: No intervention (observational study)
- Healthy: Healthy adults with no known health conditions affecting their mobility, balance, or lower extremity muscle strength
  Interventions: Other: No intervention (observational study)

INTERVENTIONS:
Other: No intervention (observational study) — No intervention; observational study

SUMMARY:
Great Toe Strength (GTS) is a potential clinical biomarker that has been associated with functional mobility and health; Additionally, GTS has been identified in the literature as one of the early symptoms of chemotherapy-induced peripheral neuropathy (CIPN). The purpose of this research study is to evaluate GTS in individuals with CIPN and healthy adults using ToeScale and see how it relates to nerve issues from chemotherapy. Additionally, we aim to assess the usability of the novel GTS assessment device, ToeScale among the participants. As a part of this study visit, you will complete some questionnaires followed by GTS and balance and gait assessments.

DETAILED DESCRIPTION:
Chemotherapy-induced peripheral neuropathy, or CIPN, is a common side effect of cancer treatment. It affects about 30-40% of people with cancer and up to 100% of those who receive chemotherapy that can harm nerves. One of the early signs of CIPN is weakness in the muscles of the great toe, which is associated with movement and balance.

Current methods used to measure the strength of the great toe muscles have several drawbacks. They are not very sensitive to changes in strength, require expensive equipment or trained professionals, and can be subjective. To address these limitations, a new portable device called ToeScale was developed. This study aims to:

1. Check if the ToeScale device is a valid measure of great toe strength (GTS) in people with CIPN and how different GTS is among age- and sex- matched healthy adults.
2. Explore the relationship between great toe strength and the severity of CIPN symptoms.
3. Assess how easy it is for participants to use the ToeScale device.

In simpler terms, this study wants to see if the new device is reliable and accurate, how well it measures GTS in people with CIPN, and whether it's easy to use.

ELIGIBILITY:
Eligibility Criteria for Chemotherapy-Induced Peripheral Neuropathy (CIPN) group:

Inclusion Criteria:

* At least 18 years of old with the ability to independently raise and low (extend or flex) the great toe
* Able to consent and complete questionnaires in English independently and have normal to corrected vision (self-reported)
* Within 3 - 6 months of starting chemotherapy and a confirmed diagnosis of CIPN using the current clinical reference standard of Nerve conduction study.

Exclusion Criteria:

* Comorbidities including but not limited to diabetes, arthritis, hypertension, thyroid disease, and heart disease, . that have been reported to be associated with the incidence of peripheral neuropathy and/or progression of CIPN.
* Toe deformities or impairments not caused by CIPN (including but not limited to hallux valgus/varus, hallux limitus, hallux rigidus, hammer toe deformity, claw toe, bunions, webbed toes)
* Self-reported impairment or impact on the strength of the foot, ankle, and/or great toe due to past medical or surgical history.

Eligibility Criteria for Healthy Control group: The participants recruited for this group will be age- and sex- matched to the CIPN group

* Inclusion Criteria:
* At least 18 years of old with the ability to independently raise and low (extend or flex) the great toe
* Able to consent and complete questionnaires in English independently and have normal to corrected vision (self-reported)
* No known health conditions that have been reported to be associated with different impairements in mobility, balance, and muscle strength (particularly in the lower extremity)

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals with CIPN and age- and sex- matched healthy controls will be recruited for this study. The recruitment will primarily rely on the resources availale through and rehabilitation specialists working within the University of Florida (UF) Health Cancer Center as well as UF Health Hospitals.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-08-05 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Great Toe Strength | Baseline
  Measured using the ToeScale, the novel device used in this study to evaluate both flexion and extension strength of the great toe
Functional Assessment of Cancer Therapy/Gynecologic Oncology Group-Neurotoxicity (FACT/GOG-Ntx) | Baseline
  This is a questionnaire that will be used to evaluate the severity of symptoms of chemotherapy-induced peripheral neuropathy (CIPN). The scores from this questionnaire will be used to conduct a deeper analysis of the differences in great toe strength within the CIPN group.
System Usability Scale (SUS) Questionnaire | Baseline
  This questionnaire will be administered at the end of the study visit, once the participants have a chance to use the device independently to evaluate their perspective on the satisfaction, ease of use, and comfort of the device.

SECONDARY OUTCOMES:
Gait analysis | Baseline
  Five trials of walking at a a self-selected pace will be conducted during which, a markerless motion capture system will be used for video data collection, that will then be used for gait analyses including spatiotemporal and kinematic variables.
Balance Assessment | Baseline
  The HUR Smart balance platform will be used to evaluate balance using two tests: The romberg test (Stable and unstable conditions) and the limits of stability test.
Timed Up and Go (TUG) | Baseline
  This is a clinical functional mobility test with a standardized protocol and measured in time (in seconds), which is currently used in clinical practice to assess fall risk. Additionally, the markerless motion capture will be used during this assessment as well to further analyze the biomechanics during different phases of the TUG assessment. We will conduct 3 trials of this assessment.
Feedback ineterview | Baseline
  This is a semi-structured interview with 7 questions that we developed based on the study protocol and assessments to obtain the participants' overall perspectives on the different aspects of the study, device, and experience. This feedback will be used for secondary thematic analyses, which will inform the development of next generation of the ToeScale as well as to improve the experience of future participants that enroll in our study. This will be the last outcome to be administered to the participants at the end of the study visit.

OTHER OUTCOMES:
Demographics Questionnaire | Baseline
  Demographic data, including age, gender, history ofathleticism, physical activity, pre-existing conditions, and medical/surgical history, will be collected before the strength and mobility assessments. This data will be used to analyze participant characteristics and potential correlations with outcome measures.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
The de-identified data might be shared with permission from the funder and PI per request and as appropriate.
Supporting Information: Study Protocol
Time Frame: After completion of study and publication of the results from the primary outcomes.
Access Criteria: Only de-identified data will be shared with permission from the funder and PI per request.
URL: https://top.ot.phhp.ufl.edu